CLINICAL TRIAL: NCT06463522
Title: Safety and Efficacy of Autologous Tumor-infiltrating Lymphocytes Therapy in Patients With Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-2024-3-48-2
Record Dates: First submitted 2024-04-26; First posted 2024-06-17 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Tumor-infiltrating Lymphocytes
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Autologous Tumor-infiltrating Lymphocytes Therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor-infiltrating Lymphocytes Therapy (Experimental): Autologous Tumor-infiltrating Lymphocytes Therapy, 2.0*10^7/Kg, single intravenous infusion.
  Interventions: Procedure: Autologous Tumor-infiltrating Lymphocytes

INTERVENTIONS:
Procedure: Autologous Tumor-infiltrating Lymphocytes — Autologous Tumor-infiltrating Lymphocytes, 2.0*10^7/Kg, single intravenous infusion.

SUMMARY:
This is a Phase 1, open label clinical trial of tumor-infiltrating lymphocytes for the treatment of patients with hepatocellular carcinoma. The purpose of this study is to assess the safety of tumor-infiltrating lymphocytes therapy in patients with hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years;
2. Diagnosis of HCC with BCLC stage B/C;
3. Anticipated survival time is longer than 3 months;
4. Liver function grade Child-Pugh A or B, without hepatic encephalopathy;
5. Left ventricular ejection fraction (LVEF) ≥ 50%;
6. ECOG physical status 0-2;
7. Laboratory tests at baseline meet the following: Absolute neutrophil count >1.0 x 109/L; Absolute neutrophil count >1.0 x 109/L; White blood cell count > 2.0 x 109/L; Platelet count > 60 x 109/L; Hgb > 8.0 g/dL; ALT and AST ≤ 5 times the upper limit of normal (ULN), Serum total bilirubin (TBiL) ≤ 51 mmol/L, or < 3 times the ULN.
8. Female subjects of childbearing potential must take acceptable measures to minimize the likelihood of pregnancy during the trial. Female subjects of childbearing potential must have a negative serum or urine pregnancy result within 48 hours prior to treatment;
9. Able to receive treatment and follow-up, including the need for the subject to receive treatment at the enrollment center.

Exclusion Criteria:

1. Pregnant or breastfeeding women;
2. WIth HIV/AIDS infection;
3. Active infection with a temperature >38.3°C prior to study treatment and have been treated with antibiotics within 2 weeks prior to enrollment;
4. Presence of the following pre-existing or concomitant diseases: Prior diagnosis of a severe autoimmune disease requiring systemic immunosuppression (steroids) for a prolonged period of time (more than 2 months), or immune-mediated symptomatic disease; Prior diagnosis of autoimmune-induced motor neuron disease; Prior toxic epidermal necrolysis release; Subjects with any psychiatric condition, including dementia, altered mental status, which may interfere with treatment in this study; Subjects with other malignancies in the previous 5 years; Subjects with heart failure ≥ grade 2 (NYHA) or hypertension uncontrolled by standard therapy; Subjects with unstable or active peptic ulcer or gastrointestinal bleeding; Subjects with serious uncontrollable disease, as determined by the study, that may interfere with treatment in this study;
5. Subjects undergoing treatment with systemic steroids;
6. Subjects who have previously used immune cell therapy (CIK, DC, DC-CIK, LAK therapy) and are less than 28 days from the end of treatment to screening;
7. Subjects who are allergic to cell therapy products or related drugs;
8. Subjects who have previously received an organ transplant or are planning to receive an organ transplant;
9. Subjects requiring anticoagulant therapy (warfarin or heparin);
10. Subjects who are judged by the investigator to be unsuitable for participation in this study due to other conditions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | day0, day3, week1, week2, week4, week12, week24
  Safety and Tolerability of Autologous Tumor-infiltrating Lymphocytes Therapy

SECONDARY OUTCOMES:
Concentration of Total Bilirubin (TBIL, mg/dL) | day0, day3, week1, week2, week4, week12, week24
  Total bilirubin refers to the concentration of bilirubin in a patient's blood sample, which is automatically measured by the laboratories in accordance with standard operating procedures.
Child-Turcotte-Pugh(CTP) score | day0, day3, week1, week2, week4, week12, week24
  CTP score is currently the most commonly used model to evaluate liver reserve function and prognosis in patients with cirrhosis. This model evaluates liver function based on HE grade, degree of abdominal fluid accumulation, bilirubin (TBiL), albumin (Alb) and prothrombin time (PT). The score ranges from 0 to 15, with the higher the score, the worse the prognosis.
Quality of life of patients | day0, day3, week1, week2, week4, week12, week24
  Quality of life assessed by Functional Assessment of Cancer Therapy - Hepatobiliary Symptom Index， which has a score ranges 0-32, a higher score indicates better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Junliang Fu, PhD, MD, Principal Investigator — the Fifth Medical Center of PLA
Locations (1):
- the Fifth Medical Center of PLA, Beijing, China